CLINICAL TRIAL: NCT07165782
Title: Brief Videos Delivered by Text Messages as a Public Health Intervention for PTSD in Youth: A Feasibility and Acceptability Randomized Trial
Brief Title: Brief Videos Delivered by Text Messages as a Public Health Intervention for PTSD in Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1031707; FDN148371 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Post-Traumatic Stress Disorder in Adolescence; Post-Traumatic Stress Disorder, PTSD; Post-Traumatic Stress Disorder in Youth
Keywords: posttraumatic stress disorder; post-traumatic stress disorder; trauma; public health; rct; text message; video intervention
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Video Intervention (Active Comparator): Participants will receive three text messages per week for 10 weeks. Each message contains a link to a video providing information about PTSD and coping strategies.
  Interventions: Behavioral: Brief Videos Delivered by Text Message
- Control Group (No Intervention): The control group will receive no intervention. They will have access to the intervention after they complete all study activities, however they will not be included in the data analysis.

INTERVENTIONS:
Behavioral: Brief Videos Delivered by Text Message — The intervention consists of brief videos delivered by text message, designed to deliver psychoeducation, coping strategies, and social support guidance for youth with PTSD. The focus is to reduce avoidance behaviors, increase exposure, change cognitions and enhance social support.
  The text messages will follow a six-module curriculum, covering key PTSD recovery topics:
  1. Psychoeducation on PTSD - Understanding symptoms, trauma responses, and brain plasticity.
  2. Reducing Avoidance - Encouraging gradual engagement with feared thoughts and situations.
  3. Cognitive Coping Strategies - Introducing cognitive restructuring techniques.
  4. Behavioral Coping Strategies - Teaching relaxation techniques (e.g., deep breathing, grounding).
  5. Social Support - Highlighting the role of social support and strategies to strengthen connections.
  6. Maintenance and Relapse Prevention - Preparing for setbacks and reinforcing progress.
  Arms: Brief Video Intervention

SUMMARY:
The goal of this clinical trial is to learn if informational videos (the intervention) sent by text messages can help young people (age 15 - 25) manage symptoms of post traumatic stress disorder (PTSD). This is a small-scale trial to evaluate whether the intervention has potential to be effective, whether it is feasible to carry out a bigger study, and whether youth find the intervention acceptable.The main questions it aims to answer are:

1. Does the intervention help youth reduce their symptoms of PTSD, anxiety, and depression, improve how well they function day-to-day, and lead to post-traumatic growth.
2. Will it be possible to conduct a larger study on the intervention (e.g., are we able to attract participants to take part in the study; do participants follow through with the intervention and the study) and is the intervention acceptable to youth (e.g., do they watch the videos, and rate the videos as useful, interesting, understandable, and relevant)?

Researchers will compare those who receive the intervention right away to those who wait to receive the intervention to see if there are differences between groups.

Videos will teach youth about PTSD and provide the opportunity to practice strategies that have been shown to help with reduce symptoms of PTSD, such as exposure, reducing avoidance, social support, and coping strategies (e.g., changing your thoughts, deep breathing, and muscle relaxation).

The study is fully online. Participants will be randomly placed in one of two groups:

1. Intervention Group: Gets three PTSD-related text messages per week for 10 weeks. They will also be asked to rate each of the videos on how helpful you found them.
2. Waitlist Group: Does not receive text messages until AFTER the final surveys for the study are completed (i.e., 5 months), then will receive the intervention.

Everyone will be asked to complete online surveys about their mental health and functioning 3 times during the study:

* Beginning of the study
* 10 weeks into the study
* 3 months after the videos end (end of study)

ELIGIBILITY:
Inclusion Criteria:

* Likely diagnosis of PTSD as indicated by a minimum score of 31 on the Post Traumatic Stress Disorder Checklist
* Direct exposure to actual or threatened death, serious injury, or sexual violence or through witnessing, learning it happened to a close relation as assessed by the Life Events Checklist
* Between 15 and 25 years old at time of enrolment
* Access to a mobile phone and a data plan that allows them to receive text messages and videos
* Live in Canada

Exclusion Criteria:

* Presence of active suicidality, determined by items from the Patient Safety Screener
* Active symptoms of psychosis, indicated by a brief Psychosis Screener Questionnaire
* An inability to read and/or understand English

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-09-10 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Posttraumatic Stress as Assessed by the PTSD Checklist (PCL-5) at 10 Weeks (End of Treatment) | From enrolment to the end of treatment at 10 weeks
  The PCL-5 is a 20-item self-report measure assessing PTSD symptom severity based on Diagnostic Statistical Manual of Mental Disorders (DSM-5) criteria. Participants rate how much symptoms have bothered them in the past month on a scale from 0 (not at all) to 4 (extremely). Symptom scores range from 0 to 80, with higher scores indicating more severe symptoms. A score of 31 or higher indicates a probable diagnosis of PTSD.

SECONDARY OUTCOMES:
Change in Posttraumatic Stress as Assessed by the PTSD Checklist (PCL-5) at 3 Months After Treatment | 3 Months After Treatment (22 weeks after enrolment)
  The PCL-5 is a 20-item self-report measure assessing PTSD symptom severity based on Diagnostic Statistical Manual of Mental Disorders (DSM-5) criteria. Participants rate how much symptoms have bothered them in the past month on a scale from 0 (not at all) to 4 (extremely). Symptom scores range from 0 to 80, with higher scores indicating more severe symptoms. A score of 31 or higher indicates a probable diagnosis of PTSD.
Change in Anxiety Score as Measured by the Generalized Anxiety Disorder-7 (GAD-7) at 10 Weeks After Enrolment (Post-Treatment) and 3 Months After Treatment | From enrolment to the end of treatment at 10 weeks and 3 months after treatment ends.
  The GAD-7 is a 7-item measure assessing generalized anxiety symptoms. Higher scores indicate greater anxiety severity.
Change in Depression Score as Measured by the Patient Health Questionnaire-9 (PHQ-9) at 10 Weeks After Enrolment (Post-Treatment) and 3 Months After Treatment | From enrolment to the end of treatment at 10 weeks and 3 months after treatment ends.
  The PHQ-9 is a 9-item measure assessing depression symptoms. Higher scores indicate greater depression severity.
Change in Functional Impairment Scores as Measured by the Sheehan Disability Scale (SDS) at 10 Weeks After Enrolment (Post-Treatment) and 3 Months After Treatment. | From enrolment to the end of treatment at 10 weeks and 3 months after treatment ends.
  The SDS will assess the severity of functional impairment. Higher scores indicate more impairment.
Change in Posttraumatic Growth as Measured by The Posttraumatic Growth Inventory - Short Form (PTGI-SF) at 10 Weeks After Enrolment and 3 Months After Treatment | From enrolment to the end of treatment at 10 weeks and 3 months after treatment ends.
  The PTGI-SF is a 10-item measure assessing positive psychological changes following trauma.

OTHER OUTCOMES:
Feasibility and Acceptability as Measured by Engagement and Video Ratings | From enrolment to end of treatment (10 weeks)
  The feasibility and acceptability of the text message-based intervention will be assessed throughout the study using recruitment and retention rates (i.e., number of participants enrolled and completing follow-ups), message engagement (i.e., number of messages rated by participants), and participant satisfaction (i.e., ratings of message helpfulness, relevance, and supportiveness). After each text, participants will be asked to rate how useful, relevant, interesting, and understandable they found the messages on a scale of 0 (not at all) to 4 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J McGrath, PhD, Principal Investigator — IWK Health
Locations (1):
- IWK Health, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes
During the informed consent process, study participants are invited to provide consent for their de-identified study data to be shared with other researchers only with the consent of the study participants. Data from those who consent may be shared with researchers provided they have ethics board approval. All participant data except for identifying data may be shared.